CLINICAL TRIAL: NCT07055373
Title: The Safety and Feasibility of Transauricular Vagus Nerve Stimulation Therapy in Chronic Whiplash-Associated Disorders: A Randomized Pilot Trial
Brief Title: Transauricular Vagus Nerve Stimulation for Chronic Whiplash Associated Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Vivo Cura Health (Other)
Responsible Party: Principal Investigator, Ashley Smith, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB25-0529
Record Dates: First submitted 2025-06-09; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Whiplash Associated Disorder (WAD)
Keywords: Whiplash Associated Disorder (WAD); Vagus Nerve Stimulation; Parasympathetic Nervous System; Sympathetic Nervous System; Post-traumatic Stress; Central Sensitization; Heart Rate Variability; Pupillometry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transauricular Vagal Nerve Stimulation (Active Comparator): Upon enrolment, participants randomized into the active treatment arm will be asked to complete a series of questionnaires seeking information on physical measurements (height, weight, & BMI), accident history, current symptoms, treatments received to date, and quality of life. Physical assessments will be performed to assess autonomic function and pain sensitivity including pupillary light reflex, heart rate variability, temporal summation, pressure pain thresholds, and conditioned pain modulation. Transauricular vagal nerve stimulation (taVNS) will be delivered a via a device that sends mild electrical pulses through the tragus of the outer ear. Participants will receive instructions device use in order to complete four weeks of twice daily (morning and evening) 45 minute sessions of taVNS. Follow ups will be completed immediately post intervention and at 4-6 weeks and 12 weeks 1 month post active taVNS. Participants will be asked to track device usage and report any adverse events.
  Interventions: Device: Transauricular Vagal Nerve Stimulation
- Sham Transauricular Vagal Nerve Stimulation (Sham Comparator): Participants assigned to the sham treatment arm will be asked to complete all the same questionnaires and physical assessments as those assigned to the active treatment arm. They will also be provided with a taVNS device and instructions on use. The device will be programed by the research team to reduce the output to '0' and thus those assigned to the sham group will not actually be receiving any active treatment. Participants will not be able to distinguish if any treatment is being received.
  Interventions: Device: Transauricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transauricular Vagal Nerve Stimulation — Transauricular VNS will be administered using the Parasym aVNT (auricular vagal neuromodulation therapy) Device (Nurosym, London, UK). The Parasym aVNT Device delivers non-invasive neuromodulation targeting the auricular branch of the vagus nerve via the tragus of the outer ear. All participants will receive four weeks of twice daily (morning and evening) 45-minute sessions of taVNS (frequency ≥ 25Hz; pulse width =250µs (Fig). The safety and tolerability of taVNS has been demonstrated in seven studies with a total of 205 (116 active, 121 sham) cardiovascular patients. Stimulation protocols ranged from 43 min to 8 hrs daily, for 1 day to 6 months. There were no device-related serious adverse events. Three patients (1.5%) experienced minor adverse events, i.e., dermal paresthesias (light tingling at the ear). No differences in tolerability were observed between active and sham taVNS [21].
  Other Names: taVNS

SUMMARY:
Approximately 50% of people with chronic whiplash-associated disorders (WAD) continue to report the presence of symptoms 12 months post-injury. These symptoms include high levels of pain and disability as well as psychological symptoms such as post-traumatic stress. The nervous system may also be affected, specifically the autonomic nervous system which is responsible for regulating heart rate and blood pressure.

An important part of the autonomic system is the vagus nerve, which helps regulate pain and stress responses. Treatment of this nerve via transauricular vagal nerve stimulation (taVNS) has been shown to improve health outcomes in many pain conditions such as chronic low back pain and postural tachycardia syndrome. TaVNS works by sending mild electrical pulses through the ear.

This project aims to explore whether or not taVNS can help people with chronic whiplash-associated disorders (WAD) feel better. The first goal is to evaluate the safety and feasibility of taVNS. The investigators are interested in learning how many people with chronic WAD participate in the study and how many complete the full treatment, as well as ensuring that the treatment does not cause any serious side effects. An additional goal is to evaluate the effects of taVNS on neck pain intensity and associated disability, pain sensitivity, heart rate variability, blood pressure, quality of life, post-traumatic stress, stress, anxiety, and depression as measured by questionnaires and physical assessments, as compared to those assigned to the sham treatment.

DETAILED DESCRIPTION:
Approximately 50% of people with chronic whiplash-associated disorders (WAD) continue to report the presence of symptoms 12 months post-injury. Many of these patients present with high levels of pain and disability and a heterogeneous presentation of both physical and psychological manifestations, inclusive of central nervous system hyperexcitability. Autonomic dysfunction has also been demonstrated in WAD.

Autonomic dysregulation via impaired peripheral vasoconstrictor responses has been demonstrated in both acute and chronic WAD, although the association with clinical features and health outcomes is unclear. Dysregulation of the hypothalamic-pituitary-adrenal axis (one of the key pathways to respond to stress) via reduced reactivity and enhanced negative feedback suppression has also been demonstrated in chronic WAD. In association with high levels of psychological distress and post-traumatic stress symptoms, stress system dysfunction in the form of autonomic nervous system (ANS) dysregulation is possible.

Previous resaerch by the investigators has demonstrated changes in autonomic function through heart rate and blood pressure measures in chronic WAD. More recently, the role of the ANS in chronic WAD has been examined using pupillometry. The results showed the presence of increased sympathetic nervous system activity, and reduced parasympathetic activity. These findings are consistent with those observed in other chronic pain conditions. This imbalance reportedly decreases the ANS adaptive response to both physical or emotional pain. These findings support the hypothesis that autonomic dysfunction potentially contributes to pain persistence.

An important link between the autonomic system and pain regulation mechanisms is the vagus nerve. Pain control occurs through vagally mediated afferent and efferent stimuli. The vagus nerve is also known to carry around 75% of parasympathetic fibers. Treatments affecting vagally mediated pain control includes non-invasive vagus nerve stimulation (VNS).

Transauricular VNS (taVNS) has been shown to improve health outcomes in many dysautonomic conditions and pain, such as chronic low back pain and postural tachycardia syndrome. Improvements in both biomarkers of autonomic dysfunction, such as heart rate variability (HRV); in association with reductions of pain and disability and improvements in pain sensitivity have been demonstrated, illustrating the potential of tVNS to modulate pain.

The specific objectives of this study are as follows:

1. The primary objective is to evaluate the safety and feasibility of a randomized pilot study of taVNS as a treatment for patients with WAD in terms of recruitment (greater than 30%), attendance (70% total treatment time in a 4 week period), retention (greater than 70% complete protocol), safety (no severe adverse events and less than a 30% increase in adverse effects for the active group), and acceptability of the protocol.
2. The secondary exploratory objectives are to evaluate neck pain intensity and associated disability, pain sensitivity, HRV, blood pressure, quality of life, post-traumatic stress, stress, anxiety, and depression - as measured by questionnaires and physical assessments - following active taVNS compared to sham taVNS in patients with WAD.

This will be a randomized, sham-controlled, participant and assessor blinded, pilot trial evaluating the safety and feasibility of taVNS for the treatment of WAD symptoms. Consenting and eligible participants will be asked to complete baseline questionnaires, physicial measurements (height, weight, and BMI), and clinical measurements. Questionnaires and physical measurements will be repeated immediately 1 month post taVNS and at 8-10 & 16 weeks. Participants will be be asked to refrain from taking prescribed medications, performing physical exercise, or consuming alcohol or coffee on day of testing. Blood pressure, heart rate variability, and pupillary light reflex measures will be performed. Participants will be instructed on use of a taVNS device including precautions and safety information.

Following study enrolment, participants will be randomized into one of two groups: active taVNS or sham taVNS. Randomization will occur via a sealed envelope where participant numbers have been sorted into active or sham taVNS by a random number generator. Participants in the sham group will be blinded using a previously established blinding method. They will undergo a 30 second ramp up period, during which, the current will be gradually increased and then the machine will reduce the waveform to 0 whilst remaining in the 'on' mode. Assessors will be blinded to the participants grouping.

Transauricular VNS will be administered using the Nurosym aVNT (auricular vagal neuromodulation therapy) Device (Parasym, London, UK). The Nurosym aVNT Device delivers non-invasive neuromodulation targeting the auricular branch of the vagus nerve via the tragus of the outer ear. All participants will receive four weeks of twice daily (morning and evening) 45-minute sessions of taVNS (frequency ≥ 25Hz; pulse width =250µs.

ELIGIBILITY:
Inclusion Criteria:

1. Symptom duration ≥3 months and <10 years; and
2. Classifiable as WAD grade I (neck pain without physical impairments) or II (neck pain & impairment such as movement loss and/or tenderness) or III (neck pain & neurological deficit evident on physical exam);
3. Average pain intensity (over one week) ≥ 4/10;
4. Neck Disability Index score > 28% (14/50).

Exclusion Criteria:

1. WAD IV injury (no neurological deficit, fracture, or dislocation);
2. Concussion symptoms;
3. Patients who have undergone cervical vagotomy;
4. Patients diagnosed with severe bradycardia;
5. Patients with a permanent implanted metallic or electronic device or jewellery at close proximity to the ear tragus;
6. Patients with any active implanted device (including electronic and/or medical devices) e.g. cochlear implant, cerebral shunts, invasive vagus nerve stimulators, or non-active but potentially interacting with the nervous system (e.g., metal implants);
7. Open wounds or rashes, swollen, red, infected, or inflamed areas or skin eruptions (e.g., phlebitis, thrombophlebitis, varicose veins); or cancerous lesions in the area of stimulation
8. Using medications associated with ANS function such as Beta Blockers;
9. Adverse general health factors such as presence of a neurological disorder (e.g., multiple sclerosis), inflammatory condition (e.g., rheumatoid arthritis), cardiovascular disorder (known severe coronary disease or recent myocardial infarction (within 5 years)); metabolic disorder (e.g., diabetes), visual deficit or disease process (e.g. cataracts, double or blurred vision), known or suspected serious spinal pathology (e.g. metastatic disease of the spine), pregnancy, or previous spinal surgery or recurrent treatment for spinal disorders;
10. History of any mental health conditions prior to the MVC, such as bipolar disorder, schizophrenia, anxiety, PTSD or severe depression;
11. People who are unable to complete the questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs); recruitment rate; attendance rate; retention rate. | The study duration is 4 months, including 1 month of self-administered taVNS. Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  The primary objective is to evaluate the safety and feasibility of a randomized pilot study of taVNS as a treatment for patients with WAD in terms of recruitment (greater than 30%), attendance (70% total treatment time in a 4 week period), retention (greater than 70% complete protocol), safety (no severe adverse events and less than a 30% increase in adverse effects for the active group), and acceptability of the protocol.

SECONDARY OUTCOMES:
Neck pain intensity as measured by the Numerical Pain Rating Scale, 0-10. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Neck pain intensity will be measured via the Numerical Pain Rating Scale (NPRS). This scale ranges from 0-10 with a higher score indicating more pain intensity.
Neck-related disability as measured by the Neck Disability Index, 0-50. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Neck-related disability will be measure by the Neck Disability Index. This test ranges betweeen a score of 0-50 with higher scores meaning increased severity of neck-related disability.
Pain sensitivity as measured by Pressure Pain Thresholds in Newtons. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Changes in pain sensitivity will be measured by assessing presure pain thresholds. An algometer will be placed on the leg or neck region and pressure will be increased until the moment when the sensation of pressure first becomes painful. At this point, the pressure will stop being applied and the value will be recorded in Newtons.
Temporal Summation as measured by NPRS, 0-10. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Temporal summation will be measured using a pin prick. The pin prick will be gently raised and lowered over the hand region, without piercing the skin, to the beat of a metronome - 1 every second. The pain will be recorded at various times at different intervals by utilizing the Numerical Pain Rating Scale (NPRS) which ranges from 0-10.
Sensitivity to pressure as measured by Conditioned Pain Modulation (% change from baseline). | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Sensitivity to pressure will be measured by Conditioned Pain Modulation (CPM). A blood pressure cuff will by worn on the upper arm and the pressure will be increased until the pain experienced is 5/10. At that time, pressure will also be applied to the shin to test the sensitivity in this region. The pressure pain threshold (PPT) on the shin will be compared before and during the arm pain from the cuff. The change in sensitivity will be recorded as a percentage of the baseline value. A lower pressure senstivity during the cuff main indicates suggests better pain tolerance. Pain inhibition is indicated if the percentage is negative.
Heart rate variability (RMSSD in ms). | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Heart rate variability (HRV) will be measured via HRV4Training app and the root mean square of successive differences (RMSSD) will be recorded in ms. RMSSD is a measure of HRV which calculats the variability of the heart rate in one minute.
Blood pressure recorded in mmHg. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Blood pressure will be recorded while seated using a standard arm cuff (sphygmomanometer).
Quality of life as measured by SF-12. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Quality of life will be evaluated using the Short Form-12 (SF-12) questionnaire which measures both a physical component summary (PCS0) and mental component summary (MCS) score. Higher scores reflect better health status.
PTSD symptoms as measured by the PCL-5. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  PTSD symptoms will be assesed using the PCL-5 questionnaire. This questionnaire consists of 20 questions reflecting DSM-5 PTSD criteria. The answer to each question is rated 0-4 with the total score ranging from 0-20. Higher scores indicated increased PTSD symptom severity.
Depression, anxiety, and stress via DASS-21. | Outcome measures will be assessed at baseline, immediately post-treatment (end of week 4) and during follow-ups at Week 8-10 and Week 16.
  Changes in depression, anxiety, and stress will be measured using the DASS-21 questionniare consisting of 21 questions measuring symptoms of each condition. Each question can be rated on a 4-point Likert scale. Scores for each of the three subscales (7 questions each) are summed and multiplied by 2 to give a final score for each condition ranging from 0-42. Higher scores indicated increased symptom severity for each condition.

OTHER OUTCOMES:
taVNS Diary | To be completed twice daily during 4 weeks of taVNS treatment.
  Daily diary for participants to track their AM and PM sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Smith, Principal Investigator — University of Calgary
Locations (1):
- Vivo Cura Health, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasylynuk C, Smith A. The Relationship Between Clinical Measures of Nociplastic Pain and Pupillary Light Reflex Measures in Chronic WAD. An observational study. 2024 IFOMPT. Basel, Switzerland2024.
- [Background] Tracy LM, Ioannou L, Baker KS, Gibson SJ, Georgiou-Karistianis N, Giummarra MJ. Meta-analytic evidence for decreased heart rate variability in chronic pain implicating parasympathetic nervous system dysregulation. Pain. 2016 Jan;157(1):7-29. doi: 10.1097/j.pain.0000000000000360. PMID 26431423
- [Background] Forte G, Troisi G, Pazzaglia M, Pascalis V, Casagrande M. Heart Rate Variability and Pain: A Systematic Review. Brain Sci. 2022 Jan 24;12(2):153. doi: 10.3390/brainsci12020153. PMID 35203917
- [Background] Koenig J, Falvay D, Clamor A, Wagner J, Jarczok MN, Ellis RJ, Weber C, Thayer JF. Pneumogastric (Vagus) Nerve Activity Indexed by Heart Rate Variability in Chronic Pain Patients Compared to Healthy Controls: A Systematic Review and Meta-Analysis. Pain Physician. 2016 Jan;19(1):E55-78. PMID 26752494
- [Background] Gockel M, Lindholm H, Niemisto L, Hurri H. Perceived disability but not pain is connected with autonomic nervous function among patients with chronic low back pain. J Rehabil Med. 2008 May;40(5):355-8. doi: 10.2340/16501977-0172. PMID 18461260
- [Background] Meints SM, Garcia RG, Schuman-Olivier Z, Datko M, Desbordes G, Cornelius M, Edwards RR, Napadow V. The Effects of Combined Respiratory-Gated Auricular Vagal Afferent Nerve Stimulation and Mindfulness Meditation for Chronic Low Back Pain: A Pilot Study. Pain Med. 2022 Aug 31;23(9):1570-1581. doi: 10.1093/pm/pnac025. PMID 35148407
- [Background] Sator-Katzenschlager SM, Scharbert G, Kozek-Langenecker SA, Szeles JC, Finster G, Schiesser AW, Heinze G, Kress HG. The short- and long-term benefit in chronic low back pain through adjuvant electrical versus manual auricular acupuncture. Anesth Analg. 2004 May;98(5):1359-64, table of contents. doi: 10.1213/01.ane.0000107941.16173.f7. PMID 15105215
- [Background] Stavrakis S, Chakraborty P, Farhat K, Whyte S, Morris L, Abideen Asad ZU, Karfonta B, Anjum J, Matlock HG, Cai X, Yu X. Noninvasive Vagus Nerve Stimulation in Postural Tachycardia Syndrome: A Randomized Clinical Trial. JACC Clin Electrophysiol. 2024 Feb;10(2):346-355. doi: 10.1016/j.jacep.2023.10.015. Epub 2023 Nov 22. PMID 37999672
- [Background] Geng D, Liu X, Wang Y, Wang J. The effect of transcutaneous auricular vagus nerve stimulation on HRV in healthy young people. PLoS One. 2022 Feb 10;17(2):e0263833. doi: 10.1371/journal.pone.0263833. eCollection 2022. PMID 35143576
- [Background] Uzlifatin Y, Arfianti L, Wardhani IL, Hidayati HB, Melaniani S. Effect of transcutaneous auricular vagus nerve stimulation in addition to exercises on disabilitiy in chronic low back pain patients: A randomized controlled study. Anaesth Pain Intensive Care 2023; 21(1):73-81.
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Spitzer WO, Skovron ML, Salmi LR, Cassidy JD, Duranceau J, Suissa S, Zeiss E. Scientific monograph of the Quebec Task Force on Whiplash-Associated Disorders: redefining "whiplash" and its management. Spine (Phila Pa 1976). 1995 Apr 15;20(8 Suppl):1S-73S. No abstract available. PMID 7604354
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics 2005;4(4):287-291.
- [Background] Luche G, Dundovic S, Stavrakis S. REPORT OF SAFETY AND TOLERABILITY OF LOW-LEVEL TRAGUS VAGAL NEUROMODULATION IN CARDIOVASCULAR PATIENTS. JACC 2024;83:13:178.
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Boonstra AM, Stewart RE, Koke AJ, Oosterwijk RF, Swaan JL, Schreurs KM, Schiphorst Preuper HR. Cut-Off Points for Mild, Moderate, and Severe Pain on the Numeric Rating Scale for Pain in Patients with Chronic Musculoskeletal Pain: Variability and Influence of Sex and Catastrophizing. Front Psychol. 2016 Sep 30;7:1466. doi: 10.3389/fpsyg.2016.01466. eCollection 2016. PMID 27746750
- [Background] Master CL, Podolak OE, Ciuffreda KJ, Metzger KB, Joshi NR, McDonald CC, Margulies SS, Grady MF, Arbogast KB. Utility of Pupillary Light Reflex Metrics as a Physiologic Biomarker for Adolescent Sport-Related Concussion. JAMA Ophthalmol. 2020 Nov 1;138(11):1135-1141. doi: 10.1001/jamaophthalmol.2020.3466. PMID 32970102
- [Background] Podolak OE, Arbogast KB, Nabin JB, Ciuffreda K, Grady M, Master CL. The use Of Pupillary Light Reflex in Concussed Athletes. Orthopaedic Journal of Sports Medicine 2020;8(4_suppl3):2325967120S00277.
- [Background] Wan AK, Rainville P, O'Leary S, Elphinston RA, Sterling M, Lariviere C, Sullivan MJL. Validation of an index of Sensitivity to Movement-Evoked Pain in patients with whiplash injuries. Pain Rep. 2018 Jun 20;3(4):e661. doi: 10.1097/PR9.0000000000000661. eCollection 2018 Jul-Aug. PMID 30123856
- [Background] Smith A, Pedler A. Conditioned pain modulation is affected by occlusion cuff conditioning stimulus intensity, but not duration. Eur J Pain. 2018 Jan;22(1):94-102. doi: 10.1002/ejp.1093. Epub 2017 Aug 14. PMID 28805288
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] Jobin K, Smith A, Campbell C, Schabrun SM, Galarneau JM, Schneider KJ, Debert CT. The safety and feasibility of transcranial direct current stimulation and exercise therapy for the treatment of cervicogenic headaches: A randomized pilot trial. Headache. 2025 May;65(5):845-862. doi: 10.1111/head.14887. Epub 2025 Jan 17. PMID 39825590
- [Background] Robinson-Papp J, George MC, Wongmek A, Nmashie A, Merlin JS, Ali Y, Epstein L, Green M, Serban S, Sheth P, Simpson DM. The Quantitative Analgesic Questionnaire: A Tool to Capture Patient-Reported Chronic Pain Medication Use. J Pain Symptom Manage. 2015 Sep;50(3):381-6. doi: 10.1016/j.jpainsymman.2015.03.013. Epub 2015 Apr 23. PMID 25912277
- [Background] Stark RG, Reitmeir P, Leidl R, Konig HH. Validity, reliability, and responsiveness of the EQ-5D in inflammatory bowel disease in Germany. Inflamm Bowel Dis. 2010 Jan;16(1):42-51. doi: 10.1002/ibd.20989. PMID 19475674
- [Background] Alhassani G, Treleaven J, Schabrun SSM. Combined transcranial and trans-spinal direct current stimulation in chronic headache: A feasibility and safety trial for a novel intervention. Hong Kong Physiother J. 2017 Feb 23;37:1-9. doi: 10.1016/j.hkpj.2016.11.001. eCollection 2017 Dec. PMID 30931040
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Hung M, Baumhauer JF, Licari FW, Voss MW, Bounsanga J, Saltzman CL. PROMIS and FAAM Minimal Clinically Important Differences in Foot and Ankle Orthopedics. Foot Ankle Int. 2019 Jan;40(1):65-73. doi: 10.1177/1071100718800304. Epub 2018 Oct 4. PMID 30282469
- [Background] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Tran N, Asad Z, Elkholey K, Scherlag BJ, Po SS, Stavrakis S. Autonomic Neuromodulation Acutely Ameliorates Left Ventricular Strain in Humans. J Cardiovasc Transl Res. 2019 Jun;12(3):221-230. doi: 10.1007/s12265-018-9853-6. Epub 2018 Dec 17. PMID 30560316
- [Background] White L, Smith AD, Farrell SF. Associations Between Resting Heart Rate, Resting Blood Pressure, Psychological Variables and Pain Processing in Chronic Whiplash-Associated Disorder: A Cross-Sectional Study. Pain Med. 2022 Oct 29;23(11):1882-1890. doi: 10.1093/pm/pnac075. PMID 35587744
- [Background] Gaab J, Baumann S, Budnoik A, Gmunder H, Hottinger N, Ehlert U. Reduced reactivity and enhanced negative feedback sensitivity of the hypothalamus-pituitary-adrenal axis in chronic whiplash-associated disorder. Pain. 2005 Dec 15;119(1-3):219-224. doi: 10.1016/j.pain.2005.10.001. Epub 2005 Nov 17. PMID 16298068
- [Background] Sterling M, Jull G, Kenardy J. Physical and psychological factors maintain long-term predictive capacity post-whiplash injury. Pain. 2006 May;122(1-2):102-8. doi: 10.1016/j.pain.2006.01.014. Epub 2006 Mar 9. PMID 16527397
- [Background] Sterling M, Jull G, Vicenzino B, Kenardy J. Sensory hypersensitivity occurs soon after whiplash injury and is associated with poor recovery. Pain. 2003 Aug;104(3):509-517. doi: 10.1016/S0304-3959(03)00078-2. PMID 12927623